CLINICAL TRIAL: NCT02401178
Title: The Role of Fillagrin Gene Mutations and FADS Genes Variation Through Its Effect on the Concentration of Polyunsaturated Fatty Acids Towards the Occurance of Atopic Dermatitis in Indonesian Infants
Brief Title: The Role of Filaggrin and FADS Genes on the Concentrations of PUFA Towards Its Effect on Atopic Dermatitis in Infants
Acronym: FLG-FADSgen
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, M.F.Conny Tanjung, MD, MD, Indonesia University
Other Study IDs: IndonesiaU
Record Dates: First submitted 2014-12-09; First posted 2015-03-27 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Atopic Dermatitis
Keywords: FLG-FADS genes variations-LCPUFA-atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat-plasma-cheeck cell
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Well baby: For cross-sectional study design:
  The dependent variables are LCPUFA composition from buccal. The independent variables are 17 SNP from FADS genes.
  For extended cross-sectional study design:
  The dependent variable is atopic dermatitis, while independent variables are:
  17 SNP; LCPUFA and FLG gene mutation

SUMMARY:
The incidence of atopic dermatitis has increased dramatically in this years. Atopic dermatitis occurs due to complex interactions between genetic and environmental factors. One of the genes that consistenly linked with AD occurences is filaggrin gene (FLG gene). Mutation on the gene can induce disruption in epidermal cytoskeleton aggregation which serves to form protein-lipid, thereby disrupting the skin permeability to water and outside particles such as allergens.8-14 Several attempts have been made to prevent the occurences and progressivity of AD, one of them is LCPUFA supplementation. Until now, the clinical and meta-analysis studies have shown inconsistent results, but LCPUFA intervention in early life gives more consistent and protective results. In this study investigators would like to know about the influence of FLG gene mutation to the occurrence of atopic dermatitis, to know the composition of LCPUFA in early life in order to see protective effects of several LCPUFA, to see the influences of FADS1 and FADS2 gene polymorphism towards LCPUFA concentration from umbilical artery and buccal swab in early life and at the time AD occurs, to know about the diet at the time of AD occurrence, and to know the role of the ratio of DHA towards AA level in the development of AD due to their antagonistic effects, and to see the interactions between FLG gene, FADS gene and LCPUFA level in the development of AD.

DETAILED DESCRIPTION:
STUDY DESIGN Cross-sectional design is used to know the role of FADS1 and FADS2 gene polymorphism in LCPUFA composition at birth (from umbilical artery and buccal swab), Extended cross-sectional designed is used to look at FLG gene mutation effect as the predictor of the emergence of atopic dermatitis, FADS1 and FADS2 gene polymorphism role in atopic dermatitis occurences, the role of DHA intake and DHA to AA ratio in preventing atopic dermatitis occurences in the first year of life.

STUDY POPULATION Target population is healthy term newborns. Affordable population is healthy term newborns in Jakarta. Study samples are healthy term newborns in Jakarta born in Primary Health Care in Kemayoran District, Central Jakarta whose parents consent to take part in this study.

METHODS Briefly, filaggrin gene mutation and FADS1 and FADS2 polymorphism will be examined from umbilical blood and LCPUFA level will be measured from umbilical artery and buccal swab in 400 newborns. The Material Transfer Agreement (MTA) from Indonesian Health Research and Development Institution (Badan Penelitian dan Pengembangan Kesehatan Republik Indonesia/LITBANGKES) will be included. Genotyping will be done by using iPLEX Gold chemistry (Sequenom) and MALDI-TOF (matrix assisted laser desorption ionization-time of flight) as the methods to detect allele differences.

Every month, breastfeeding; each duration of breastfeeding; formula intake; how much and what kind of formula given, if any (regular formula, hypoallergenic formula); will be monitored. At the time complementary feeding to breast milk starts, dietary analysis by Food Frequency Questionnaire (FFQ), and monitoring of body weight, length, head circumference and skin condition will be done.

If parents complain about the presence of skin disorders or there is a suspicion of AD occurfence, investigator's team will ask and accompany parents and subject to Dermatologist. If subject can not come, a home visit will be done, and photograph will be taken. The dermatologist will later confirm the diagnosis through the photo. LCPUFA level measurement will be done once more through buccal swab at the time atopic dermatitis occurs or at the end of the monitoring for subjects who do not acquire AD.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn: term, healthy, weighs more than 2500 gram, and has no congenital disorders
2. Mother : consents to take part in the study and signs the informed consent
3. Mother with normal gestational history without any complications such as gestational hypertension, gestational diabetes mellitus, not a vegetarian
4. Mother does not suffer severe illness during or after labor period
5. Mother does not get omega-3 and omega-6 supplementation during pregnancy and breastfeeding period

Exclusion Criteria:

1. Mother : gets omega-3 or omega-6 supplementation
2. Newborn: gets omega-3 or omega-6 supplementation

Ages: 1 Hour to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Target population is healthy term newborns. Affordable population is healthy term newborns in Jakarta. Study samples are healthy term newborns in Jakarta born in Primary Health Care in Kemayoran District, Central Jakarta whose parents consent to take part in this study.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of atopic dermatitis in patients with FLG gene mutation, FADS1 or FADS2 gene polymorphisms | one year
  Incidence of atopic dermatitis

SECONDARY OUTCOMES:
Association of FLG gene and atopic dermatitis | One year
  Odds ratio of FLG gene and atopic dermatitis
Association of LCPUFA composition and atopic dermatitis: | One year
  Odds ratio of LCPUFA composition and atopic dermatitis:
Analysis of genetic variation association of FADS1 & FADS2 over the level of LCPUFA | one year
  Regression coefficient and determinant coefficient to see the association between the genetic variation of FADS1 to FADS3 genes over the change of LCPUFA composition
Influence of several risk factors with atopic dermatitis | one year
  Survival analysis to see the influence of several risk factors with atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Conny F Tanjung, MD, Principal Investigator — Indonesia University
Locations (1):
- Puskesmas Kemayoran (Primary Health Care in Kemayoran District), Jakarta Pusat, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Derived] Tanjung C, Rzehak P, Sudoyo H, Mansyur M, Munasir Z, Immanuel S, Irawan R, Reischl E, Demmelmair H, Hadinegoro SR, Sjarif DR, Koletzko B. The association of fatty acid desaturase gene polymorphisms on long-chain polyunsaturated fatty acid composition in Indonesian infants. Am J Clin Nutr. 2018 Nov 1;108(5):1135-1144. doi: 10.1093/ajcn/nqy166. PMID 30475958